CLINICAL TRIAL: NCT07069257
Title: Effectiveness of Neuromuscular Electrical Stimulation Added to Oral Motor Therapy in Children With Cerebral Palsy Experiencing Drooling Problems: A Randomized Controlled Trial
Brief Title: Effectiveness of Neuromuscular Electrical Stimulation Added to Oral Motor Therapy in Cerebral Palsy
Acronym: NOMES-CP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aslinur Keles Ercisli, MD, PhD (Other)
Collaborators: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor-Investigator, Aslinur Keles Ercisli, MD, PhD, Investigator, Fatih Sultan Mehmet Training and Research Hospital
Organization: Fatih Sultan Mehmet Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-SP-SC-NMESOMT-01; Ethics Committee No: 1295 (20- (Other: Ethics Committee of Istanbul Medipol University)
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy (CP); Drooling
Keywords: Cerebral Palsy; Drooling; Sialorrhea; Oral Motor Therapy; Neuromuscular Electrical Stimulation; Pediatric Rehabilitation; Ultrasound; Masseter Muscle; Orbicularis Oris Muscle
MeSH Terms: conditions — Cerebral Palsy; Sialorrhea

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to three parallel groups: (1) oral motor therapy plus neuromuscular electrical stimulation (NMES), (2) oral motor therapy alone, and (3) oral motor therapy plus sham NMES.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blinded to group assignment. The clinician performing ultrasound assessments is also blinded. The therapist delivering the interventions and administering the scales is not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral Motor Therapy Plus NMES (Experimental): Participants assigned to this arm will receive oral motor therapy combined with active neuromuscular electrical stimulation (NMES) applied to the masseter and orbicularis oris muscles.
  Interventions: Behavioral: Oral Motor Therapy; Device: Neuromuscular Electrical Stimulation (NMES)
- Oral Motor Therapy (Other): Participants assigned to this arm will receive oral motor therapy without any NMES. This is a behavioral therapy.
  Interventions: Behavioral: Oral Motor Therapy
- Oral Motor Therapy Plus Sham NMES (Sham Comparator): Participants assigned to this arm will receive oral motor therapy combined with sham NMES that does not deliver active stimulation.
  Interventions: Behavioral: Oral Motor Therapy; Device: Sham Neuromuscular Electrical Stimulation (Sham NMES)

INTERVENTIONS:
Behavioral: Oral Motor Therapy — Structured oral motor exercises will be applied to the lips, tongue, cheeks, and jaw. Facial massage and thermal stimulation (warm and cold) will be performed. Intraoral sensory stimulation will be applied using a brush, lemon juice, and a cold metal probe.
Device: Neuromuscular Electrical Stimulation (NMES) — Active NMES will be applied bilaterally to the masseter muscles and to the orbicularis oris muscle in addition to oral motor therapy sessions, using a Chattanooga NMES device. Each application will be performed in cycles of 5 seconds of stimulation and 10 seconds of rest. The stimulation parameters will be set to a frequency of 10-15 Hz and a pulse width of 300 microseconds. The current intensity will be gradually increased to a level just above the motor threshold, sufficient to elicit a noticeable pulling sensation without causing discomfort, and will be adjusted according to each participant's tolerance. NMES will be delivered for a total duration of 15 minutes per session. For the electrical stimulation of the orbicularis oris muscle, a pen-type electrode will be used. In this procedure, four regions of the orbicularis oris muscle (upper, lower, right, and left) will be stimulated in two cycles of 45 pulses each.
  Arms: Oral Motor Therapy Plus NMES
Device: Sham Neuromuscular Electrical Stimulation (Sham NMES) — Simulated neuromuscular electrical stimulation will be applied without delivering active electrical current after oral motor therapy sessions to mimic the treatment experience without producing physiological effects.
  Arms: Oral Motor Therapy Plus Sham NMES

SUMMARY:
This randomized, controlled, single-blind trial aims to investigate the effectiveness of neuromuscular electrical stimulation (NMES) combined with oral motor therapy in reducing drooling severity among children with cerebral palsy. Participants will be allocated to an intervention group (oral motor therapy plus NMES), a control group (oral motor therapy alone) and a sham group (oral motor therapy with placebo NMES).

DETAILED DESCRIPTION:
Drooling is a common and disabling problem in children with cerebral palsy, adversely affecting health, social participation, and quality of life. Oral motor therapy is frequently used to improve oral control, and neuromuscular electrical stimulation (NMES) has been suggested as an adjunctive treatment to enhance orofacial muscle function.

This randomized, controlled, single-blind study will include children aged 4 to 17 years diagnosed with cerebral palsy and presenting with moderate to severe drooling (Drooling Severity and Frequency Scale score ≥3). Participants will be randomly assigned to one of three groups: oral motor therapy alone, oral motor therapy plus active NMES, and oral motor therapy with sham NMES. The intervention comprises twelve therapy sessions over four weeks, delivered by a trained therapist.

Oral motor therapy involves exercises targeting lips, tongue, cheeks, and jaw, in addition to thermal and tactile stimulation (using brushes, spoons, cold packs, and heat packs). NMES will be applied bilaterally to the masseter muscles and to the orbicularis oris muscle using a Chattanooga NMES device. Sham NMES will simulate the procedure without delivering active stimulation.

Outcome measures will be assessed before and after the intervention and will include both subjective and objective drooling scales: Drooling Severity and Frequency Scale (DSFS), Drooling Impact Scale (DIS), Visual Analog Scale for drooling severity, Drooling Quotient (DQ5), and caregiver reports of bib usage. Orofacial muscle thickness will be measured with ultrasound imaging. Additional assessments will include functional classification systems (GMFCS, MACS, CFCS, VFCS, EDACS, FOIS) and the Pediatric Eating Assessment Tool (PEDI EAT-10).

This study is approved by the Ethics Committee of Istanbul Medipol University.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy (unilateral/bilateral spastic, ataxic, dyskinetic, or mixed type)
* Presence of drooling control problems
* Age between 4 and 17 years
* Gross Motor Function Classification System (GMFCS) levels 2, 3, 4, or 5
* Stable drooling severity for at least one month prior to enrollment
* Drooling Severity and Frequency Scale (DSFS) score of 3 or higher

Exclusion Criteria:

* Diagnosis of dysphagia
* Use of medications affecting drooling within the past 72 hours
* Upper respiratory tract infection and/or salivary gland infection during the study period
* History of botulinum toxin injection to the salivary glands

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Drooling Severity and Frequency Scale (DSFS) Score | At Baseline and at 4th Week (after completion of 12 therapy sessions)
  The Drooling Severity and Frequency Scale (DSFS) is a validated clinical tool that assesses drooling in two domains: severity and frequency.
  Severity is rated on a 5-point scale from 1 (dry; never drools) to 5 (profuse; clothing, hands, tray, and objects wet).
  Frequency is rated on a 4-point scale from 1 (never) to 4 (constantly). Higher scores in each subscale indicate more severe and frequent drooling. The total score reflects the combined impact of both dimensions.
Change in Drooling Impact Scale (DIS) Score | At Baseline and at 4th Week (after completion of 12 therapy sessions)
  The Drooling Impact Scale (DIS) assesses the impact of drooling on daily life. It consists of 10 items, each scored from 1 (barely) to 10 (extremely), resulting in a total score range of 10 to 100. Higher scores indicate a greater negative impact of drooling on quality of life.

SECONDARY OUTCOMES:
Change in Orofacial Muscle Thickness Measured by Ultrasound | At Baseline and at 4th Week (after completion of 12 therapy sessions)
  Ultrasound measurement of masseter and orbicularis oris muscle thickness to evaluate changes in muscle structure following intervention.
Change in Visual Analog Scale (VAS) Drooling Severity Score | At Baseline and at 4th Week (after completion of 12 therapy sessions)
  Participants or caregivers rate the perceived severity of drooling using a 10 cm visual analog scale (VAS), ranging from 0 (no drooling) to 10 (extremely severe drooling). Higher scores indicate greater severity of drooling. The VAS is a widely used subjective assessment tool in clinical settings.
Change in Drooling Quotient (DQ5) | At Baseline and at 4th Week (after completion of 12 therapy sessions)
  The Drooling Quotient (DQ5) is an observational measure used to quantify the frequency of drooling in individuals with drooling disorders. Observations are conducted during two separate 5-minute periods: one during rest (passive state) and one during activity (active state such as talking or playing).
  During each 5-minute period, the presence or absence of drooling is recorded every 15 seconds, for a total of 20 intervals per condition. The DQ5 is calculated as the percentage of intervals in which drooling is observed (e.g., drooling observed in 6 out of 20 intervals = 30%). Higher percentages indicate more frequent drooling. Scores from both rest and activity conditions are reported.
Change in Karaduman Chewing Performance Scale (KCPS) Score | At Baseline and at 4th Week (after completion of 12 therapy sessions)
  The Karaduman Chewing Performance Scale (KCPS) evaluates chewing function in children with cerebral palsy, scored from Level 1 (normal chewing) to Level 4 (severely impaired chewing).
Change in Tongue Thrust Rating Scale (TTRS) Score | At Baseline and at 4th Week (after completion of 12 therapy sessions)
  The Tongue Thrust Rating Scale (TTRS) is a clinician-rated observational tool used to assess the severity of tongue thrust during swallowing. It is scored on a 3-point scale:
  1. = No tongue thrust,
  2. = Mild; tongue positioned between the teeth,
  3. = Moderate; tongue positioned between the lips. Higher scores indicate more pronounced tongue thrust behavior during swallowing.
Change in Daily Number of Wet Bibs and Cloths | At Baseline and at 4th Week (after completion of 12 therapy sessions)
  The total number of bibs and cloths used daily due to drooling, recorded by caregivers. Higher counts reflect increased drooling severity.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Aycan, Principal Investigator — Health Sciences University Fatih Sultan Mehmet Training and Research Hospital; Esra Giray, Assoc. Prof., Study Chair — Istanbul University of Health Sciences, Fatih Sultan Mehmet Training and Research Hospital; Aslinur Keles Ercisli, MD, PhD, Study Director — Istanbul University of Health Sciences, Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Ataşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to confidentiality concerns and institutional data sharing policies.

REFERENCES:
- [Background] Assoratgoon I, Shiraishi N, Tagaino R, Ogawa T, Sasaki K. Sensory neuromuscular electrical stimulation for dysphagia rehabilitation: A literature review. J Oral Rehabil. 2023 Feb;50(2):157-164. doi: 10.1111/joor.13391. Epub 2022 Nov 28. PMID 36357332
- [Background] Sigan SN, Uzunhan TA, Aydinli N, Eraslan E, Ekici B, Caliskan M. Effects of oral motor therapy in children with cerebral palsy. Ann Indian Acad Neurol. 2013 Jul;16(3):342-6. doi: 10.4103/0972-2327.116923. PMID 24101813
- [Background] 2. Awan, W. A., Aftab, A., Janua, U. I., Ramzan, R., & Khan, N. (2017). EFFECTIVENESS OF KINESIO TAPING WITH OROMOTOR EXERCISES IN IMPROVING DROOLING AMONG CHILDREN WITH CEREBRAL PALSY: soi: 21-2017/re-trjvol01iss02p21. The Rehabilitation Journal, 1(02), 21-27.
- [Background] 1. Fatima et al (2019), Study of the effectiveness of oromotor exercises to reduce drooling in cerebral palsy children